CLINICAL TRIAL: NCT01233037
Title: Observational Study Assessing Markers of Endothelial Function and Exercise CapaciTy in Patients With Left Ventricular Assist Devices
Brief Title: Markers of Endothelial Function and Exercise CapaciTy in Patients With Left Ventricular Assist Devices (EFECT LVAD)
Acronym: EFECT-LVAD
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1007M86679
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Endothelial Cells; Exercise Tolerance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Some of the blood collected at each visit will stored by the investigator for up to 5 years. Samples will be kept in our laboratory for up to 5 years as plasma, after which they will be destroyed. Samples will be identified only by a code number, only the principal investigator and his research staff will have access to the code. The results of the future tests will not be communicated to subjects in this study.
  The samples are stored in the form of plasma from Peripheral blood for additional markers of endothelial function (Soluble thrombomodulin, IL-6, etc.)
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a non-randomized feasibility study of endothelial function, exercise capacity, and outcome following pre-left ventricular assist device (LVAD)therapy and cardiac transplant.

The study period will be 5 years, with 20 patients to be enrolled. The investigators anticipate that 15 patients will survive to complete the one year follow up period.(the published survival rate of LVAD is 75% in one year). 10 patients are anticipated to undergo cardiac transplant within 3 years of initial enrollment and they are followed until their 2nd annual post transplant invasive evaluation.

Markers of endothelial function will be studied to permit comparison with selected clinical outcomes. The hypothesis is that the endothelial functions will be altered after implantation of LVAD then before its implantation, both acutely and chronically, and this may affect the exercise capacity, quality of life and occurrence of cardiac allograft vasculopathy post cardiac transplantation.

DETAILED DESCRIPTION:
This is a non-randomized, feasibility study of endothelial function, exercise capacity, and outcome following pre-LVAD patients through LVAD therapy and cardiac transplantation.

The study period will be 5 years. It is anticipated that 20 patients will be enrolled and 15 will survive (published survival estimate following LVAD is approximately 75% at one year) to complete the one-year follow-up period. 10 patients are anticipated to undergo heart transplant within 3 years of initial enrollment and they will be followed until their 2nd annual post-transplant invasive evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Advanced heart failure and scheduled LVAD implantation for standard clinical indications.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

* Inability to personally provide informed consent
* Medical activity restriction that precludes ambulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the University of Minnesota Cardiology Practice prior to clinically-indicated LVAD implantation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Determine which markers of vascular function are most highly associated with exercise capacity following LVAD implantation. | 3 years

SECONDARY OUTCOMES:
Determine which markers are associated with Survival following LVAD | 3 years
To determine which markers are associated with Risk of GI bleeding thought to arise from intestinal AVMs | 3 years
Determine which markers are associated with Risk and severity of coronary allograft vasculopathy at 1 and 2 years post transplant | 5 years
Determine which markers are associated with quality of life | 5 years
Obtain pilot data on the acute endothelial response to exercise in patients with LVAD | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Eckman, MD, Principal Investigator — University of Minnesota
Locations (1):
- Fairview Health Systems Research, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Tominaga R, Smith W, Massiello A, Harasaki H, Golding LA. Chronic nonpulsatile blood flow. II. Hemodynamic responses to progressive exercise in calves with chronic nonpulsatile biventricular bypass. J Thorac Cardiovasc Surg. 1996 Apr;111(4):857-62. doi: 10.1016/s0022-5223(96)70347-1. PMID 8614147
- See also: the study sponsor website — http://umn.edu
- See also: the study location — http://www.fairview.org/